CLINICAL TRIAL: NCT04572113
Title: Comparison of Cervical Motion Restriction and Interface Pressure Between Two Cervical Collars
Status: Completed | Type: Observational
Sponsor: More Foundation (Other)
Collaborators: DJO LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: 4029
Record Dates: First submitted 2020-09-13; First posted 2020-10-01 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2020-09

CONDITIONS: Cervical Pain
Keywords: Neck pain; Cervical collar
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | US Export: Yes

GROUPS / COHORTS (3):
- No collar: Cervical range of motion and tissue interface pressure measurements are recorded while subject are not wearing a cervical collar
- DJO collar: Cervical range of motion and tissue interface pressure measurements are recorded while subject are wearing a DJO cervical collar
  Interventions: Device: Cervical collar
- Miami J collar: Cervical range of motion and tissue interface pressure measurements are recorded while subject are wearing a Miami J cervical collar
  Interventions: Device: Cervical collar

INTERVENTIONS:
Device: Cervical collar — Data will be recorded while patients are not wearing or wearing one of two cervical collars
  Groups: DJO collar; Miami J collar

SUMMARY:
Cervical orthoses are used to restrict motion for the purpose of preventing spinal instability following trauma or pre- and post-surgery or to protect from pain. Modern cervical orthoses are able to effectively restrict motion of the head however load is concentrated on areas of occipital tissue and may, with long term wear, lead to tissue breakdown in the form of pressure ulcers. Previous research has shown that the Miami J collar (Össur Americas Foothill Ranch, CA) effectively reduced cervical movement while providing superior pressure relief. As new cervical orthoses are developed and become commercially available it is useful to examine their performance in comparison to existing well-tested devices. DJO Global (Vista, CA) have recently developed a cervical collar. The purpose of this study is to compare the ability of this newly developed collar to restrict cervical range of motion while at the same time limit the tissue interface pressure exerted by the collar on patients when they are in an upright seated or supine position Data will be collected in a fully equipped 3D motion analysis laboratory. Cervical range of motion will be tracked and analyzed. Interface pressures between the head and collar will be measured using custom pressure mats.

ELIGIBILITY:
Inclusion Criteria:

* English speaking.
* Subjects who have read and signed IRB approved informed consent for this study.

Exclusion Criteria:

* History of neck pain or neck injury requiring medical care within the previous 12 months.
* History of spinal surgery, physical or chiropractic therapy of the neck.
* History of cervical spondylosis or osteoporosis.
* Pregnant.
* Currently Incarcerated

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Subjects will be recruited by word of mouth from the surrounding general population and may include staff of MORE Foundation and The CORE Institute.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-01-09 (Actual); Study Completion 2019-11-02 (Actual)

PRIMARY OUTCOMES:
Cervical range of motion | At enrollment
  The subjects will be seated in a backed chair and monitored to ensure their spine remains in contact with the backrest throughout the CROM assessment. Each subject will be instructed to perform a sequence of of neck flexion-extension, lateral flexion, and rotation movements. Each movement will be repeated six times until the motion is stopped by muscle tightness, discomfort or a substitution movement occurs, without a collar, and with each study collar chosen chosen in random order. Angular range of motion in degrees will be recorded in each plane. Flexion-extension - angle between maximum flexion and maximum extension. Lateral flexion - angle between maximum right lateral flexion and maximum left lateral flexion. Rotation - angle between maximum right rotation and maximum left rotation.
Tissue interface pressure | At enrollment
  With the subject seated, 3, 75 x 120mm pressure sensor pads, each pad each consisting of 40 individual sensors; will be placed over the anterior mandibles and occiput. The subject will be fit with an appropriately sized collar. The order of collar wear will be the same as for the CROM measurements. Pressure measurements and distribution of pressure will be recorded for a period of 30 seconds. The subject will then be placed in a supine position on a standard examination table without a pillow and pressure measurements and distribution of pressure will be collected for a period of 30 seconds while the subject maintains his/her head in a relaxed position.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Jacofsky, PhD, Study Director — More Foundation
Locations (1):
- MORE Foundation, Phoenix, Arizona, United States